CLINICAL TRIAL: NCT03748381
Title: Comparison of Visual Performance of 2 Diffractive Trifocal Intraocular Lenses: a Randomised Controlled Trial
Brief Title: Comparison of 2 Diffractive Trifocal IOLs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Trifocal
Record Dates: First submitted 2018-11-19; First posted 2018-11-20 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Cataract
Keywords: Cataract surgery; Trifocal IOL
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trifocal IOL (Experimental): The patients will receive two different diffractive trifocal IOLs in each eye (AT Lisa tri vs. Rayner trifocal) during cataract surgery
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery — During cataract surgery patients will be implanted with the AT Zeiss Lisa tri in one eye and the Rayner trifocal in the contralateral eye

SUMMARY:
Compare two commercially available bilateral implanted diffractive trifocal lenses (Zeiss AT Lisa tri vs. Rayner trifocal) after cataract surgery concerning visual function and spectacle independence.

DETAILED DESCRIPTION:
Spectacle independence is a central aim in modern cataract surgery. Although bilateral monofocal IOL implantation, aiming for emmetropia or low myopia, leads to high levels of patient satisfaction in distance vision, spectacle dependence for reading and other near vision tasks is the usual result.

The option commonly used to achieve spectacle independence are multifocal intraocular lenses (IOLs). Multifocal IOLs either use a refractive or diffractive design or a combination of both or segmented asymmetric optics. The principal of the refractive design is based on changing the route of light rays by thickness, curvature and optical density of the lens. The principal of diffractive design is based on scattering of light rays when passing an edge in the material of the lens. One potentially negative aspect of multifocal refractive IOLs is pupil size dependence, another is loss of light energy to higher order diffraction which is not useful to the patient. In clinical studies diffractive lenses resulted in a better outcome in terms of optical quality, better contrast sensitivity and lens photopic phenomena (dysphotopsia such as halos and glare) than in refractive lenses.

Until recently multifocal lenses were typically bifocal with a focus assigned to near and a focus assigned to far vision. However, the intermediate working distance is poorly covered by that multifocal design. Since objects commonly viewed in this distance include computer displays and tablets, the intermediate distance has become a crucial part in daily life. As a consequence of poor intermediate visual acuity there is a need for spectacles for intermediate vision. Variations in the addition of power chosen for near vision provided some intermediate visual acuity but still suboptimal.

Therefore, a new concept of multifocality has been recently introduced, i.e. the trifocal lens. Trifocal lenses provide three focal distances, far, intermediate and near. This ideally results in even less spectacle dependence, including computer work. There are currently 3 trifocal designs available and are being used readily. One potential disadvantage of trifocal compared to bifocal IOLs is that near vision may be slightly poorer with the need for reading glasses with prolonged fine near work.

A slightly modified trifocal design has been recently introduced, that appears to have even better near vision than other trifocal designs as well as the potential for less dysphotopsia with a dilated pupil such as during the night.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract
* Scheduled for bilateral cataract extraction
* Motivated to be less spectacle dependant
* Age 21 and older
* Corneal astigmatism ≤ 1.5 D (Keratometry, IOL Master 700)
* written informed consent prior to recruitment

Exclusion Criteria:

* Pregnancy (pregnancy test will be taken pre-operatively in women of reproductive age)
* Retinitis pigmentosa
* Chronic uveitis
* Amblyopia
* Pupil decentration > 1mm center shift
* preceded retinal surgery
* preceded Laser-in-situ-Keratomileusis (LASIK)
* Any ophthalmic abnormality that could compromise visual function or the measurements

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Uncorrected Near Visual Acuity | 12 months
  Uncorrected Near Visual Acuity will be assessed with ETDRS charts

SECONDARY OUTCOMES:
Uncorrected and Best corrected Far and Intermediate Visual Acuity, | 12 months
  Uncorrected and Best corrected Far and Intermediate Visual Acuity will be assessed with ETDRS charts
Halo measurements | 12 months
  Halos will be assessed using the Halometer App on a tablet
Reading speed | 12 months
  Reading speed will be assessed using the Salzburg Reading Desk
Defocus curve | 12 months
  A defocus curve will be done by adding glasses starting from -4.0D to +2.0D to the best corrected far correction
Contrast sensitivity | 12 months
  Contrast sensitivity will be assessed using the Optec Vision tester

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided